CLINICAL TRIAL: NCT05765617
Title: Effect Of Calcitriol On Neutrophil To Lymphocytes Ratio And High Sensitivity C-Reactive Protein Covid-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, M.D., Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAP03
Record Dates: First submitted 2023-03-09; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: calcitriol, HsCRP
MeSH Terms: conditions — COVID-19 | interventions — Calcitriol

STUDY DESIGN:
Intervention Model Description: This research was an observational analytic cohort retrospective study in which the subjects were moderate degree COVID-19 inpatients in Sebelas Maret University Hospital divided into two groups. The control group received standard therapy, while the treatment group received calcitriol 2x400 iu per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study used calcitriol and a placebo, which were similar in shape; researchers and patients did not know who was getting the drug or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo 2x1 per day
  Interventions: Other: Placebo
- Calcitriol (Experimental): the treatment group received calcitriol 2x400 iu per day for 5 day
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol — The treatment group received calcitriol 2x400 iu per day for five days. Calcitriol uses Oscal, obtained from Kalbe Pharma
  Other Names: Oscal
  Arms: Calcitriol
Other: Placebo — Placebo give 2x1 per day for five day
  Arms: Control

SUMMARY:
This research is a study that compares the administration of calcitriol with the outcomes of COVID-19 patients

DETAILED DESCRIPTION:
This research was an observational analytic cohort retrospective study in which the subjects were moderate degree COVID-19 inpatients in Sebelas Maret University Hospital divided into two groups. The control group received standard therapy, while the treatment group received calcitriol 2x400 iu per day.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients, hospitalized patients, and patients aged 18-60 years

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
HsCRP | Hs CRP (high sensitive c reactive protein) examination was carried out on the first day of hospitalization and the 5th day of hospitalization
  High-sensitivity C-reactive protein (hsCRP) is a marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Universitas Sebelas Maret Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No